CLINICAL TRIAL: NCT00382538
Title: A Randomized, Placebo-Controlled, Double-Blinded Study of Mifepristone in Midtrimester Termination of Pregnancy
Brief Title: Mifepristone and Mid-Trimester Termination of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24597
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Abortion, Induced; Abortion, Second Trimester
Keywords: mifepristone; induction; abortion; injection, intra-amniotic

INTERVENTIONS:
Drug: Addition of mifepristone 200 mg 24 hours before induction

SUMMARY:
Mid-second trimester medical terminations of pregnancy require admission to the hospital for the length of time it takes a woman to abort. The current protocol at BMC uses intra-amniotic digoxin injection the day prior to admission. The following day, the woman is admitted and given sequential doses of misoprostol until delivery occurs. The average length of time between the first dose of misoprostol and delivery is 12 hours, requiring most women to stay overnight. This is a randomized, placebo-controlled, double-blinded study designed to determine whether adding mifepristone significantly reduces the induction interval time (time between starting the first misoprostol and delivery) required for a second trimester termination.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blinded study.

Allocation Method: Women will be randomized using a computer-run random number table. Tablets will be placed in capsules by the pharmacy according to the randomization chart.

Blinding: Subjects will receive a capsule containing either 200 mg of mifepristone or 250 mg Vitamin C. Neither she nor the researcher will be aware of which medication she receives.

Outcomes: The primary outcome measured will be the mean interval from first misoprostol dose to fetal expulsion. Secondary outcomes include the proportion of women delivering within 24 hours from the first dose of misoprostol and the proportion of women with a complete delivery not requiring additional treatment for retained placenta. We will also compare the amount of pain medication used, as well as the length of hospital stay between the two groups.

Inclusion criteria Inclusion criteria: · Need for second trimester induction for termination of pregnancy · Gestational age of 18-23 weeks · At least 18 years of age or 16 years old with parental consent No medical contraindication to the use of digoxin and misoprostol for the purposes of inducing abortion. · Able and willing to give informed consent in English or Spanish

Exclusion criteria Exclusion criteria: · Known allergy to mifepristone, misoprostol or prostaglandins · Pre-existing intrauterine fetal demise · Premature preterm rupture of membranes · IUD in place · History of chronic adrenal failure, porphyrias; or concurrent long-term corticosteroid treatment Unable or unwilling to give informed consent in English or Spanish

Involvement in the study will be as follows: on study day number one, all patients undergo an ultrasound-guided amniocentesis with intra-amniotic injection of digoxin regardless of entry into the study. Study patients will be randomized to the treatment or placebo group, and will receive one of two similar-looking tablets containing the allocated medication. The tablet will be swallowed in the clinic. The patient, researchers and the care providers will be blinded to group assignment. All patients return to the hospital the the day after their digoxin injection for induction. From this point on, the treatment of women enrolled and those not enrolled in the study will be identical; they are admitted to the hospital and induction for termination is begun using an initial 400mcg of misoprostol buccally. The initial dose is followed by 200 mcg of misoprostol every six hours until delivery is successful or 24 hours passes without delivery. Less than 5% of women require more than 24 hours of induction, and approximately 15% require extraction of the placenta if it does not pass spontaneously after the fetus. The subjects enrolled will not differ from other termination patients in regards to the following: 1. the number of appointments or time required in the hospital 2. use of intra-amniotic digoxin 3. termination method; misoprostol, 400 mg, followed by 200 mg every 6 hours 4. pain medication administration (PCA narcotics) 5. Medical evaluation of need to use other methods of completing abortion if 24 hours has elapsed after first misoprostol dose without delivery.

Analytic Plan:

The primary outcome is the length of induction interval for termination. The Kaplan-Meier procedure will be utilized to create a survival curve for analysis of induction to delivery interval by time. Demographic data for each group will also be compared to assure that there are no other differences between groups. Chi -square analysis will be used for dichotomous variables and t-tests for continuous variables.Study Size and Power:

A power calculation was performed for time from induction to delivery using a significant value of 0.05 and power of 80% using a survival analysis power formula. We used our previous data to estimate the mean time of induction and then estimated a likely delta (difference between the two treatment groups) of 35%. The number of patients needed in each group using this calculation is 32, and therefore the total number needed is 64.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or over
* able to give informed consent in English or Spanish
* Requesting termination of pregnancy

Exclusion Criteria:

* Under 16 years of age
* rupture membranes or intrauterine death

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64
Dates: Start 2005-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Time from start of induction to fetal delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Borgatta, MD, MPH, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kapp N, Borgatta L, Stubblefield P, Vragovic O, Moreno N. Mifepristone in second-trimester medical abortion: a randomized controlled trial. Obstet Gynecol. 2007 Dec;110(6):1304-10. doi: 10.1097/01.AOG.0000289577.32274.a5. PMID 18055725